CLINICAL TRIAL: NCT02348255
Title: A Phase II, Multi-institutional Trial of NOVO-TTF-100A, BCNU and Bevacizumab for GBM in First Relapse
Brief Title: NovoTTF-100A With Bevacizumab and Carmustine in Treating Patients With Glioblastoma Multiforme in First Relapse
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor Accrual
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH); NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC#249; 663113 (Other: UC Davis); UCDCC#249 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH); NCI-2014-02628 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Adult Brain Glioblastoma; Recurrent Adult Brain Neoplasm
MeSH Terms: conditions — Brain Neoplasms | interventions — Bevacizumab; Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (bevacizumab, carmustine, NovoTTF-100A) (Experimental): Patients receive bevacizumab IV over 30-90 minutes every 2 weeks beginning on day -7 for up to 13 doses and carmustine IV over 4 hours every 8 weeks beginning on day 1 for up to 3 doses. Patients also undergo NovoTTF-100A according to standard procedures starting one week before the first dose of carmustine.
  Interventions: Procedure: Electric Field Therapy; Biological: Bevacizumab; Drug: Carmustine; Other: Quality-of-Life Assessment

INTERVENTIONS:
Procedure: Electric Field Therapy — Undergo NovoTTF-100A
Biological: Bevacizumab — Given IV
  Other Names: Avastin; rhuMab-VEGF
Drug: Carmustine — Given IV
  Other Names: FDA 0345
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trial studies the safety of NovoTTF-100A in combination with bevacizumab and carmustine and to see how well they work in treating patients with glioblastoma multiforme that has returned for the first time. NovoTTF-100A, a type of electric field therapy, delivers low intensity, alternating "wave-like" electric fields that may interfere with multiplication of the glioblastoma multiforme cells. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as carmustine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving NovoTTF-100A together with bevacizumab and carmustine may be an effective treatment for glioblastoma multiforme.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Establish the safety of NovoTTF-100A in combination with bevacizumab and BCNU (carmustine) in glioblastoma multiforme (GBM) patients who have relapsed after chemoradiation therapy (first relapse).

II. Determine the 6 month overall survival (OS). III. Determine the 6 month progression free survival (PFS). IV. Evaluate the effect of this therapy regimen on quality-of-life.

OUTLINE:

Patients receive bevacizumab intravenously (IV) over 30-90 minutes every 2 weeks beginning on day -7 for up to 13 doses and carmustine IV over 4 hours every 8 weeks beginning on day 1 for up to 3 doses. Patients also undergo NovoTTF-100A according to standard procedures starting one week before the first dose of carmustine.

After completion of study treatment, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed GBM
* Progressive disease after temozolomide and radiation therapy (in "first relapse")
* At least 28 days since chemotherapy or radiation
* Karnofsky performance score at least 70%
* Platelet count >= 130/mm^3
* Absolute neutrophil count >= 1500/mm^3
* Calculated creatinine clearance greater than 45 mg/dl using the Cockcroft-Gault formula
* Aspartate aminotransferase (AST) < 2 times the upper limit of normal
* Bilirubin < 1.5 times the upper limit of normal
* Subjects with child-bearing potential agree to use effective means of contraception

Exclusion Criteria:

* Prior systemically administered nitrosoureas or vascular endothelial growth factor (VEGF) targeted therapy
* Chemotherapy for glioma other than temozolomide or Gliadel wafers (steroids are allowed)
* Pregnant or breast feeding
* Active inflammatory bowel disease
* Abdominal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months
* Hypertension: systolic blood pressure (SBP) > 150 or diastolic blood pressure (DBP) > 100 mm mercury (Hg) despite antihypertensive medications
* New York Heart Association (NYHA) grade II or greater congestive heart failure (CHF); myocardial infarction or unstable angina within 6 months
* History of thrombosis
* Symptomatic peripheral vascular disease, stroke or transient ischemic attack within 6 months
* Bleeding risks: Required to be on therapeutic anticoagulation (aspirin is allowed), coagulopathy (e.g. hemophilia or von Willebrand's disease); any grade III or greater hemorrhage, major surgical procedure, or significant trauma within 28 days; core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days
* Activated partial thromboplastin time (APTT) must not exceed 32.5 seconds (normal range 21.8-31.5 seconds); international normalized ratio (INR) must not exceed 1.30 (normal range 0.87-1.18)
* Serious, non-healing wound, ulcer, or bone fracture
* Active implanted medical device (e.g. deep brain stimulators, spinal cord stimulators, vagus nerve stimulators, pacemakers, defibrillators, and programmable shunts), a skull defect (such as missing bone with no replacement), a shunt, or bullet fragments
* Known sensitivity to conductive hydrogels like the gel used on electrocardiogram (ECG) stickers or transcutaneous electrical nerve stimulation (TENS) electrodes
* Human immunodeficiency virus (HIV) positive
* Proteinuria at screening as demonstrated by urine dipstick >= 2+
* Prior organ transplantation
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Aspirin, nonsteroidal anti-inflammatory drugs (NSAIDs), clopidogrel or any other drug whose goal is to inhibit platelet function
* Unable to give signed informed consent

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events, assessed by National Cancer Institute-Common Terminology Criteria 4.0 toxicity criteria | Up to 12 months
  Toxicity summaries will be provided for all subjects who have received any part of the study treatment. Statistical analysis will include estimates of proportions with each class of toxicity with a 95% confidence interval.
Progression Free Survival | Time from first day of treatment to the first observation of disease progression or death due to any cause, assessed up to 6 months
  Will be estimated using the product-limit method of Kaplan and Meier.
Overall Survival | Time from first day of treatment to time of death due to any cause, assessed up to 6 months
  Will be estimated using the product-limit method of Kaplan and Meier.
Quality of life as measured using the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 and BN-20 brain cancer module | Up to 6 months
Change in tumor volume using magnetic resonance imaging (MRI) | Baseline to day 168
  Mean change in linear dimension will be evaluated for shrinkage using a paired t-test. If the assumption of normality is violated, a signed rank test will be used. The Response Assessment in Neuro-oncology (RANO) criteria will be part of the MRI evaluation.
Change in linear dimension using MRI | Baseline to day 168
  Mean change in linear dimension will be evaluated for shrinkage using a paired t-test. If the assumption of normality is violated, a signed rank test will be used. The RANO criteria will be part of the MRI evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Robert O'Donnell, Principal Investigator — University of California, Davis
Locations (2):
- United States (2):
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Piedmont Hospital, Atlanta, Georgia